CLINICAL TRIAL: NCT01352884
Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of AMP-224 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMP-224-01
Record Dates: First submitted 2011-05-06; First posted 2011-05-12 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Cancer
Keywords: Cancer; Carcinoma; Tumor; Solid tumor; Metastatic; Melanoma
MeSH Terms: conditions — Neoplasms; Carcinoma; Neoplasm Metastasis; Melanoma

ARMS (2):
- Stage 1 (Experimental): Stage 1 will identify the recommended Stage 2 dose using a dose-escalation process. Dose-escalation will continue until either a maximum tolerated dose is established, or a therapeutic dose is reached.
  Interventions: Drug: AMP-224
- Stage 2 (Experimental): Stage 2 will further explore the safety, pharmacokinetics, and preliminary clinical activity of AMP-224 in at least one tumor type based on pharmacodynamic assessments and clinical activity emerging from the Dose-Escalation Phase. Tumor tissue and blood specimens will be evaluated for pharmacodynamic markers/activity at specified timepoints throughout the study.
  Interventions: Drug: AMP-224

INTERVENTIONS:
Drug: AMP-224 — Escalating doses of AMP-224
  Arms: Stage 1
Drug: AMP-224 — Stage 2 will further explore the safety, pharmacokinetics, and preliminary clinical activity of AMP-224 in at least one tumor type based on pharmacodynamic assessments and clinical activity emerging from the Dose-Escalation Phase. Tumor tissue and blood
  Arms: Stage 2

SUMMARY:
This is a Phase 1, open-label, multi-center, first time in human study of AMP-224 in adult patients with cancer that is not responding to standard therapy. This study will be conducted in two stages consisting of a Dose-Escalation stage and an Expansion Stage.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide informed consent
* In Dose-Escalation: Must have solid tumor malignancy or cutaneous T-cell lymphoma that has relapsed and is refractory to standard therapy, or for which no standard therapy exists
* In Expansion Phase: Must have melanoma or ovarian cancer that is histologically or cytologically confirmed
* Ovarian cancer patients must have recurrent of persistent non-mucinous disease, and must not have received more than 2 prior chemotherapeutic regimens
* Melanoma patients must have recurrent or persistent non-ocular AJCC Stage IIIC or IV disease that is surgically incurable and unresectable
* Melanoma patients with documented BRAF mutation that is known to be responsive to BRAF inhibitors must have failed or be intolerant to such inhibitors
* Must have measurable disease
* Must be able to provide access to archival (Dose-Escalation Phase) and/or fresh tumor tissue (Dose-Escalation and Expansion Phases) at Screening prior to study entry
* Must by at least 18 years old
* Must have adequate organ function

Exclusion Criteria:

* Prior cancer therapies must have completed at least 14 days or 5 half-lives (whichever is longer) prior to first dose of AMP-224
* Prior treatment with an anti-PD1 antibody therapy
* Known antibody response against prior antibody therapy or fusion protein therapeutics
* Major surgery within 4 weeks prior to first dose of AMP-224
* Prior allogeneic or autologous bone marrow or organ transplantation
* Known and/or a history or evidence of autoimmune disease except vitiligo, resolved childhood asthma and stable hypothyroidism
* Received an immunomodulatory drug within 2 weeks of first dose of AMP-224
* Active infections requiring antibiotics, physician monitoring, or recurrent fevers >100.4 degrees fahrenheit associated with a clinical diagnosis of active infection
* Patients with cirrhosis
* Clinically significant cardiac or electrocardiogram abnormalities
* History or evidence of HIV
* Active viral disease (except when the viral infection is associated with the malignancy)
* Regular use of illicit drugs or a recent history of substance abuse
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events. | From start of study drug administration until the date of first documented progression or date of death from any cause; through Day 56 of final cycle.
Number of participants with dose-limiting toxicities. | From start of study drug administration until the date of first documented progression or date of death from any cause: through Day 56 of the final cycle.
Number of participants with changes in laboratory values, vital signs, physical exam, and electrocardiogram. | From start of study drug administration until the date of first documented progression or date of death from any cause: through Day 56 of the final cycle.
Determine Maximum Tolerated Dose based on the occurrence of dose-limiting toxicities. | From start of study drug administration through Day 28 of Cycle 1.
Determine Recommended Phase 2 Dose following analysis of adverse events, pharmacokinetics and changes in laboratory evaluations. | From start of study drug administration until withdrawal; through Day 56 of final cycle.

SECONDARY OUTCOMES:
Evaluate pharmacokinetics, including area under the plasma concentration versus time curve (AUC), peak plasma concentration (Cmax) and clearance of AMP-224 following single and repeat doses of AMP-224. | From Day 0 pre-dose through Day 56 of final cycle.
Evaluate Overall Response Rate (ORR), including Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progression-Free Survival (PFS). | From Screening through 12 weeks following final cycle.
Characterization of the effects of AMP-224 on its receptor, PD-1, in peripheral T cells via flow cytometry and correlate with response to treatment. | From Screening until 12 weeks post-final cycle.
Evaluation and correlation between response to treatment and expression of PD-1 on tumor infiltrating T cells or in available malignant pleural effusions via flow cytometry and/or immunohistochemistry. | Screening through 12 weeks post-final cycle.
Evaluation and correlation between response to treatment and expression of B7-H1 on tumors via immunohistochemistry. | Screening through 12 weeks post-final cycle.
Identification of peripheral patient selection and pharmacodynamic markers from blood samples that predict and/or correlate with response to treatment. | Screening through 12 weeks post-final cycle.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- [Derived] Borch TH, Donia M, Andersen MH, Svane IM. Reorienting the immune system in the treatment of cancer by using anti-PD-1 and anti-PD-L1 antibodies. Drug Discov Today. 2015 Sep;20(9):1127-34. doi: 10.1016/j.drudis.2015.07.003. Epub 2015 Jul 17. PMID 26189934